CLINICAL TRIAL: NCT00000965
Title: Pharmacokinetics of Total Phosphorylated Zidovudine in Mononuclear Cells From HIV-Infected Patients
Brief Title: The Effects of Zidovudine on the Blood of HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Purpose: Treatment
Other Study IDs: ACTG 161
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Leukocytes, Mononuclear; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Phosphorylation
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To define the pharmacokinetic parameters (blood levels) of total phosphorylated zidovudine (AZT) in peripheral blood mononuclear cells (PBMC) from HIV-infected patients.

Despite an understanding of the serum (or plasma) pharmacokinetics (blood levels) of AZT, a therapeutic concentration range and optimal dosing interval have not yet been determined.

DETAILED DESCRIPTION:
Despite an understanding of the serum (or plasma) pharmacokinetics (blood levels) of AZT, a therapeutic concentration range and optimal dosing interval have not yet been determined.

Three studies are planned on two separate patient groups. Group (1) Patients who have never taken AZT start on a standard dose of AZT. Blood samples are taken hourly for an 8-hour period on days 1 and 14. Other blood samples are taken on days 2, 4, and 8. Group (2) Patients who have never taken AZT are given a standard dose for the first week, increasing each week until week 5. Blood samples are taken at the end of each weekly treatment. After 4 weeks of standard treatment, patients in groups 1 and 2 return and receive a single morning dose of oral AZT. Blood samples are taken immediately before dosing and at 1, 2, 4, 6, and 8 hours after dosing. After a 48-hour clearance period, patients return and resume dosing. Blood samples are again taken over an 8-hour period. After 24 weeks of standard treatment, the pharmacokinetic studies are repeated.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* FDA-approved anti-pneumocystis and antifungal prophylactic or suppressive regimens.
* Acyclovir for up to 3 weeks intermittently.

Patients must:

* Meet current guidelines for receiving prescription zidovudine.
* Have written informed consent from both subject and parent or guardian if under 18. Be capable of understanding and giving informed consent. Women and minorities are actively encouraged to participate.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malabsorption syndrome (3 or more loose stools/day for at least 4 weeks associated with unintentional weight loss of greater than 10 percent of body weight).

Concurrent Medication:

Excluded:

* Probenecid or non-FDA approved investigational drugs.
* Systemic chemotherapy.
* Other antiviral agents, licensed or investigational, including ganciclovir, foscarnet, ribavirin, didanosine (ddI), dideoxycytidine (ddC), and dideoxydidehydrothymidine (D4T).

Chronic acyclovir.

-

Patients with the following are excluded:

* Active bacterial, fungal, or viral infection requiring systemic therapy not specifically allowed.
* Significant, chronic medical conditions that could impair compliance with study treatment.

Prior Medication:

Excluded:

* Zidovudine (AZT).
* Systemic chemotherapy within previous 6 months.
* Acyclovir within 30 days of study entry.

Risk Behavior:

Excluded:

* Unable to take oral medication reliably.
* Alcohol or drug abuse that could impair compliance with study treatment.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Primary Completion 1993-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B Stretcher, Study Chair; P Frame, Study Chair; A Pesce, Study Chair
Locations (1):
- Univ of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Stretcher BN, Pesce AJ, Frame PT, Greenberg KA, Stein DS. Correlates of zidovudine phosphorylation with markers of HIV disease progression and drug toxicity. AIDS. 1994 Jun;8(6):763-9. doi: 10.1097/00002030-199406000-00007. PMID 8086134
- [Background] Stretcher BN. Pharmacokinetic optimisation of antiretroviral therapy in patients with HIV infection. Clin Pharmacokinet. 1995 Jul;29(1):46-65. doi: 10.2165/00003088-199529010-00006. PMID 7586898
- [Background] Stretcher BN, Pesce AJ, Frame PT, Stein DS. Pharmacokinetics of zidovudine phosphorylation in peripheral blood mononuclear cells from patients infected with human immunodeficiency virus. Antimicrob Agents Chemother. 1994 Jul;38(7):1541-7. doi: 10.1128/AAC.38.7.1541. PMID 7979286